CLINICAL TRIAL: NCT06498336
Title: Specific miRNA Associated With Endothelial Dysfunction and Mitochondrial Damage in Patients With Septic Acute Kidney Injury
Brief Title: miRNA in Septic Acute Kidney Injury
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: University Hospital Olomouc (Other)
Responsible Party: Sponsor
Other Study IDs: INT-01-sepsis-miRNA; RVO-FNOs/2024 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2024-06-27; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Sepsis; Acute Kidney Injury; Acute Kidney Injury Due to Sepsis
Keywords: acute kidney injury; endothelial dysfunction; mitochondrial damage; Pentraxin 3; miRNA; sepsis; uromodulin
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Critically ill adult septic patients without acute kidney injury: The patients in this group will be screened clinically and by standard laboratory biochemical methods to determine sepsis diagnosis according to SEPSIS 3 (1). Blood samples for obtaining serum/plasma of the patients will be taken on the 1st and 4th day of sepsis diagnosis.
  Interventions: Diagnostic Test: Laboratory examination to determine the presence of sepsis
- Critically ill adult septic patients with acute kidney injury: The patients will be screened clinically and by standard laboratory biochemical methods to determine sepsis diagnosis according to SEPSIS 3 and acute kidney injury according to KDIGO 2012 (2). Blood samples for obtaining serum/plasma of the patients will be taken on the 1st and 4th day of sepsis diagnosis.
  Interventions: Diagnostic Test: Laboratory examination to determine the presence of sepsis and acute kidney injury
- Healthy volunteers: The blood samples for miRNA and biochemical parameters will be collected once, after randomization.
  Interventions: Diagnostic Test: Laboratory examination to determine miRNA and biochemical parameters

INTERVENTIONS:
Diagnostic Test: Laboratory examination to determine the presence of sepsis — Standard laboratory biochemical methods will be used to determine sepsis diagnosis accord-ing to SEPSIS 3 (1). Blood samples for obtaining serum/plasma of the patients will be taken on the 1st and 4th day of sepsis diagnosis.
  Groups: Critically ill adult septic patients without acute kidney injury
Diagnostic Test: Laboratory examination to determine the presence of sepsis and acute kidney injury — Standard laboratory biochemical methods will be used to determine sepsis diagnosis according to SEPSIS 3 and acute kidney injury according to Guidelines Kidney Disease Improving Global Outcomes (KDIGO) 2012 (2). Blood samples for obtaining serum/plasma of the patients will be taken on the 1st and 4th day of sepsis diagnosis.
  Groups: Critically ill adult septic patients with acute kidney injury
Diagnostic Test: Laboratory examination to determine miRNA and biochemical parameters — Laboratory examination will be performed to determine miRNA and biochemical parameters.
  Groups: Healthy volunteers

SUMMARY:
Acute kidney injury is a common and serious complication of sepsis and septic shock, which may be associated with a worse outcome of the patient's condition. The exact pathophysiological mechanism of septic acute kidney injury remains a challenge. One of the possible causes appears to be endothelial dysfunction and mitochondrial damage of renal tubular cells. The aim of this study is to identify specific microRNAs associated with these pathophysiological events in sepsis and septic acute kidney injury. And to establish a new potential diagnostic or therapeutic target for the prevention or treatment of septic acute kidney injury.

DETAILED DESCRIPTION:
Sepsis is generally characterized as a life-threatening organ dysfunction and dysregulating host reaction to the infection (e.g., bacterial, viral, mycotic (1). Typical pathophysiological processes of sepsis include systemic inflammation, immune suppression, activation of the clotting cascade, and increase of endothelial vascular permeability with subsequent leak of fluids into the interstitial space. One of the most important organ damage due to ongoing sepsis is acute kidney injury (AKI), which is also a predictor of mortality in critically ill patients. The exact pathophysiology of septic AKI remains a challenging and poorly understood mechanism. A decrease of oxygen delivery to the tissues during the septic shock and usually high oxygen consumption of renal tubular cells make them prone to ischemia injury with consequences in tubular cell death. Among potential immune inflammatory response biomarkers in sepsis and septic shock might be promising pentraxin 3 (PTX3), which plays an important role in endothelial dysfunction with several pathogenic pathways' activation. Recently has been shown the positive effect of PTX3 on the inhibition of reactive oxygen species, mitochondrial injury, and apoptosis pathway in AKI (3,4). Another promising urinary or serum biomarker of AKI seems to be uromodulin, which is dynamically regulated in response to sepsis. Serum uromodulin concentrations decrease during septic human AKI development and are associated with increased renal and systemic oxidative damage (5,6,7). MicroRNAs are small non-coding RNAs, that have been reported to be useful biomarkers for AKI development or potential target for AKI treatment. Determination of serum PTX3 and uromodulin concomitantly with specific circulating miRNAs associated with PTX3 and uromodulin-specific signaling pathways in critically ill septic patients could bring new insights to septic AKI pathophysiology and contribute to future development of new preventive or therapeutic options in septic patients.

ELIGIBILITY:
Inclusion Criteria:

The study group of patients with sepsis with or without acute kidney injury

* age > 18 years
* newly diagnosed sepsis or septic shock with or without acute kidney injury

Healthy volunteers

* no evidence of infection on clinical or laboratory examination
* age > 18 years
* signed informed consent

Exclusion Criteria:

The study group of patients with sepsis with or without acute kidney injury

* age < 18 years
* chronic kidney disease at stage 4 or 5 according to KDIGO recommendations (KDIGO) for chronic kidney disease 2024
* patients on chronic dialysis treatment, or after renal transplantation

Healthy volunteers

* acute or chronic infection
* renal disease

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients suffering from sepsis defined according to SEPSIS 3 definition, with or without acute kidney injury defined by KDIGO 2012 (2) and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Determination of serum expression of pentraxin 3 (PTX3) and uromodulin | 4 days
  To determine the concentration of serum PTX3 and serum uromodulin in critically ill septic patients and their comparison to serum concentrations of creatinine and the acute kidney injury (AKI) stage as well as to the concentrations of procalcitonin (PCT) and interleukin-6 (IL-6) as inflammation markers on day 1 and 4 of study. The serum concentrations of PTX3 and uromodulin in ng/mL will be determined also in healthy volunteers to establish the laboratory reference ranges (values).
Determination of expression and 4 days course investigation of miRNAs | 4 days
  To determine the expression and 4-day time course investigation of 7 specific circulating miRNAs associated with sepsis and septic acute kidney injury from 352 miRNA targets using a two-tailed Quantitative reverse transcription polymerase chain reaction (RT-qPCR). All selected miRNAs will be determined also in healthy volunteers to establish the laboratory reference ranges (values).
Target genes of miRNAs and their association with endothelial dysfunction and mitochondrial injury in sepsis | 4 days
  To match the target genes (from miRNA database) of these specifically expressed miRNAs with biochemical pathways associated with serum PTX3 and uromodulin involved in endothelial dysfunction of renal microvasculature, the influence of mitochondrial injury/dysfunction with reactive oxygen species production and activation of cell apoptosis in septic acute kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Naděžda Petejová, Assoc.Prof.,MD,PhD,MSc, Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Olomouc, Olomouc, Olomouc Region

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Chen J, Matzuk MM, Zhou XJ, Lu CY. Endothelial pentraxin 3 contributes to murine ischemic acute kidney injury. Kidney Int. 2012 Dec;82(11):1195-207. doi: 10.1038/ki.2012.268. Epub 2012 Aug 15. PMID 22895517
- [Background] Lee HH, Kim SY, Na JC, Yoon YE, Han WK. Exogenous pentraxin-3 inhibits the reactive oxygen species-mitochondrial and apoptosis pathway in acute kidney injury. PLoS One. 2018 Apr 19;13(4):e0195758. doi: 10.1371/journal.pone.0195758. eCollection 2018. PMID 29672566
- [Background] El-Achkar TM, Wu XR, Rauchman M, McCracken R, Kiefer S, Dagher PC. Tamm-Horsfall protein protects the kidney from ischemic injury by decreasing inflammation and altering TLR4 expression. Am J Physiol Renal Physiol. 2008 Aug;295(2):F534-44. doi: 10.1152/ajprenal.00083.2008. Epub 2008 May 21. PMID 18495803
- [Background] LaFavers KA, Hage CA, Gaur V, Micanovic R, Hato T, Khan S, Winfree S, Doshi S, Moorthi RN, Twigg H, Wu XR, Dagher PC, Srour EF, El-Achkar TM. The kidney protects against sepsis by producing systemic uromodulin. Am J Physiol Renal Physiol. 2022 Aug 1;323(2):F212-F226. doi: 10.1152/ajprenal.00146.2022. Epub 2022 Jun 27. PMID 35759740
- [Background] LaFavers KA, Macedo E, Garimella PS, Lima C, Khan S, Myslinski J, McClintick J, Witzmann FA, Winfree S, Phillips CL, Hato T, Dagher PC, Wu XR, El-Achkar TM, Micanovic R. Circulating uromodulin inhibits systemic oxidative stress by inactivating the TRPM2 channel. Sci Transl Med. 2019 Oct 2;11(512):eaaw3639. doi: 10.1126/scitranslmed.aaw3639. PMID 31578243
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD Work Group. KDIGO 2024 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease. Kidney Int. 2024 Apr;105(4S):S117-S314. doi: 10.1016/j.kint.2023.10.018. No abstract available. PMID 38490803
- See also: 2. Kidney Disease Improving Global Outcomes (KDIGO) Acute Kidney Injury Work Group. KDIGO Clinical Practice Guideline for Acute Kidney Injury. Kidney inter., Suppl. 2012; 2: 1-138. — https://kdigo.org